CLINICAL TRIAL: NCT02445066
Title: A Pilot Study to Examine the Effects of Vitamin D Supplementation on Mitochondrial Bioenergetics in Older Adults - An EVIDENCE Sub-Study
Brief Title: A Pilot Study to Examine the Effects of Vitamin D Supplementation on Mitochondrial Bioenergetics in Older Adults
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00028235
Record Dates: First submitted 2015-05-11; First posted 2015-05-15 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Low 25-hydroxyvitamin D Concentrations
Keywords: Vitamin D
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open label (Other): Vitamin D3 - 4,000 IU/day for 4 months
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3

SUMMARY:
This pilot study is a 4-month open label trial in 15 older (65-89 yrs) men and women with initial 25(OH)D concentrations of 12-<18 ng/mL to explore the effect of increasing 25(OH)D concentrations to ≥30 ng/mL through vitamin D3 supplementation on changes in mitochondrial bioenergetics. We will assess the bioenergetic profile of blood cells isolated mitochondria, and muscle fibers as well as the expression of mitochondrial proteins and regulators of mitochondria biogenesis before and after supplementation. All participants will be given vitamin D3 (4,000 IU/d) for 4 months.

DETAILED DESCRIPTION:
In the past two decades, the role of vitamin D has extended beyond bone health to encompass a wide range of biological activities important to muscle function in older adults. Low 25-hydroxyvitamin D (25[OH]D) concentrations (<30 ng/mL) are associated with lower extremity muscle weakness, impaired physical performance, and slower walking speed,(1-8) known risk factors for disability.(9-15) Low 25(OH)D concentrations in older adults have also been associated with frailty as well as the individual frailty components including muscle weakness, slow walking speed, and exhaustion/fatigue.(16-18) Clinical findings of vitamin D deficiency (25(OH)D <12 ng/mL) include proximal muscle weakness, muscle pain, and gait impairments which are often reversed with vitamin D supplementation.(19;20) However, vitamin D's effects on the mechanisms underlying muscle function are not well understood. Recent evidence supports a role for vitamin D in skeletal muscle mitochondrial metabolism. Using 31P-MRS imaging, an increase in maximal mitochondrial oxidative phosphorylation (OXPHOS) has been reported following vitamin D supplementation.(21) Thus, we hypothesize that muscle weakness and slow walking speed in individuals with low 25(OH)D concentrations may in part be due to diminished OXPHOS activity and lower ATP generation in skeletal muscle mitochondria.

Vitamin D insufficiency is common in older adults, ranging from approximately one-third to three-fourths of community-dwelling adults aged ≥70 years depending on the cut-point used (25(OH)D <20 ng/mL or <30 ng/mL, respectively).(22;23) Similarly, bioenergetic decline is broadly associated with increasing age.(24) Thus, examining the association between vitamin D and mitochondrial bioenergetics can improve our understanding of the underlying mechanisms and range of potential benefits of remediating low 25(OH)D concentrations in older adults.

The objective of the study is to obtain preliminary data on the effect of increasing 25(OH)D concentrations among older adults with vitamin D insufficiency to ≥30 ng/mL through vitamin D3 supplementation on 1) bioenergetic profiles of multiple blood cell populations, skeletal muscle mitochondria, and muscle fibers and 2) skeletal muscle mitochondrial mass and biogenesis.

Hypothesis 1: Bioenergetic capacity as well as respiratory control in muscle mitochondria, muscle fibers, and blood cells will be improved following 4 months of vitamin D3 supplementation.

Hypothesis 2: Expression of key mitochondrial proteins (VDAC/Porin and COX4) and regulators of mitochondria biogenesis (PGC1a, SIRT1, SIRT3, and TFAM) will be higher following 4 months of vitamin D3 supplementation.

We plan to recruit individuals only from screen fails of the EVIDENCE study (IRB00022395). The EVIDENCE study is enrolling 200 participants whose 25(OH)D concentrations are 18-<30 ng/mL. Those whose concentrations are 12-<18 ng/mL at their EVIDENCE screening visit will be approached about participating in this pilot study. We will utilize the EVIDENCE screen fails because this is a pilot study with limited funding, the screening labs (25(OH)D) are expensive and the number needed to screen would be cost-prohibitive in a pilot study, and these two studies are run in the same clinic with the same staff. All screening measures will occur during the EVIDENCE study and measures will begin for this study at the baseline visit.

All persons who screen fail for EVIDENCE with a 25(OH)D concentration of 12-<18 ng/mL will be informed that they are not eligible for the EVIDENCE study and will be called with these results. If they meet all of the same eligibility criteria for this study which eliminates participants with conditions that may affect their ability to safely perform the neuromuscular function tests, consume vitamin D supplements, or undergo a muscle biopsy, these people will be informed that we have another study for those whose vitamin D levels are insufficient. If interested, they will be asked to come in for a baseline visit (as long as this visit can occur within 2 months of their EVIDENCE screening visit). Those persons who screened more than 2 months ago for the EVIDENCE study will not be eligible for this study as the lab work and other tests performed may no longer be accurate.

ELIGIBILITY:
Inclusion Criteria:

* SPPB score of 10 or less
* initial serum 25(OH)D concentration of 12-17.9 ng/mL
* not dependent on a walker
* willing to provide informed consent and to adhere to the protocol
* not involved in another behavioral, exercise, or investigational drug intervention study
* self-reported physical performance difficulty
* were screened for the EVIDENCE study within the last 2 months

Exclusion Criteria:

* serious or uncontrolled chronic disease
* evidence of impaired cognitive function (MoCA<18)
* taking prescription vitamin D2 or taking >1000 IU/day of vitamin D3 from all sources; taking an oral corticosteroid; taking hormone replacement therapy
* inability or contraindications to consume daily vitamin D supplements
* knee or hip surgery within the last 6 months or planned knee or hip surgery within the next year
* not willing or eligible to undergo a muscle biopsy (on blood thinners)
* weight loss of greater than or equal to 5% in the past 3 months
* BMI > 40kg/m2
* eye surgery within the past month or planned within the next month
* if the PI feels the participant is unlikely to follow the protocol

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Respirometric profiling | 4 months
  Respirometry of isolated mitochondria will be performed in order to examine intrinsic mitochondrial function (type1). Respirometry of permeabilized muscle fibers will be performed to assess type 2 alterations in mitochondrial function. Mitochondrial mass and biogenesis will be determined by western blot analysis. Blood based bioenergetic profiling - PBMC's, monocytes, lymphocytes, and platelets will be separated from whole blood and assessed for basal respiration, maximal respiration, ATP linked respiration, spare respiratory capacity, proton leak, and non-mitochondrial respiration.

SECONDARY OUTCOMES:
Lower extremity muscle power | 4 months
  The Nottingham Power Rig will be used for assessing power output from the lower limbs. Participants sit in a chair and unilaterally depress a foot lever, which is attached to a flywheel, as hard and as fast as they can. Power output, derived from the acceleration of the flywheel, will be recorded in Watts.
Physical performance | 4 months
  Physical performance will be assessed using the expanded Short Physical Performance Battery, the Timed Up and Go tests, and Usual and Fast walking speeds over 20 meters.
Grip strength | 4 months
  Grip strength will be measured using an isometric hydraulic hand dynamometer (Jamar, Bolingbrook, IL)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Molina, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States